CLINICAL TRIAL: NCT04405076
Title: A Phase 2a, Randomized, Observer-Blind, Placebo Controlled, Dose-Confirmation Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1273 SARS-COV-2 Vaccine in Adults Aged 18 Years and Older
Brief Title: Dose-Confirmation Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1273 COVID-19 Vaccine in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1273-P201; 75A50120C00034 (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2020-05-13; First posted 2020-05-28 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; mRNA-1273.351; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID 19; COVID 19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A is observer-blind. During Part B participants may request to be unblinded by scheduling a Participant Decision clinic visit. Part C is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- mRNA-1273: Dose 50 microgram (ug) - Participants Aged 18-54 years (Experimental): Part A: Participants aged 18-54 years will receive 1 intramuscular (IM) injection of 50 ug mRNA-1273 on Day 1 and on Day 29.
  Part B: Participants aged 18-54 years who choose to be unblinded and received 50 ug mRNA-1273 during Part A, will receive 1 IM injection of mRNA-1273 (booster dose) on Day 1.
  Interventions: Biological: Biological: mRNA-1273
- mRNA-1273: Dose 50 ug - Participants Aged 55+ years (Experimental): Part A: Participants aged 55+ years will receive 1 IM injection of 50 ug mRNA-1273 on Day 1 and on Day 29.
  Part B: Participants aged 55+ years who choose to be unblinded and received 50 ug mRNA-1273 during Part A, will receive 1 IM injection of mRNA-1273 (booster dose) on Day 1.
  Interventions: Biological: Biological: mRNA-1273
- mRNA-1273: Dose 100 ug - Participants Aged 18-54 years (Experimental): Part A: Participants aged 18-54 years will receive 1 IM injection of 100 ug mRNA-1273 on Day 1 and on Day 29.
  Part B: Participants aged 18-54 years who choose to be unblinded and received 100 ug mRNA-1273 during Part A, will receive 1 IM injection of mRNA-1273 (booster dose) on Day 1.
  Interventions: Biological: Biological: mRNA-1273
- mRNA-1273: Dose 100 ug - Participants Aged 55+ years (Experimental): Part A: Participants aged 55+ years will receive 1 IM injection of 100 ug mRNA-1273 on Day 1 and on Day 29.
  Part B: Participants aged 55+ years who choose to be unblinded and received 100 ug mRNA-1273 during Part A, will receive 1 IM injection of mRNA-1273 (booster dose) on Day 1.
  Interventions: Biological: Biological: mRNA-1273
- Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 18-54 years (Placebo Comparator): Part A: Participants aged 18-54 years will receive 1 IM injection of mRNA-1273-matching placebo on Day 1 and on Day 29.
  Part B: Participants aged 18-54 who choose to be unblinded and received mRNA-1273-matching placebo during Part A, will receive 1 IM injection of 100 ug mRNA-1273 on Day 1 and Day 29.
  Interventions: Biological: Biological: mRNA-1273; Biological: Placebo
- Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 55+ years (Placebo Comparator): Part A: Participants aged 55+ years will receive 1 IM injection of mRNA-1273-matching placebo on Day 1 and on Day 29.
  Part B: Participants aged 55+ years who choose to be unblinded and received mRNA-1273-matching placebo during Part A, will receive 1 IM injection of 100 ug mRNA-1273 on Day 1 and Day 29.
  Interventions: Biological: Biological: mRNA-1273; Biological: Placebo
- mRNA 1273.351 20 ug (Part C) (Experimental): Part C: Participants will receive 1 IM booster dose of 20 ug of mRNA 1273.351 on Day 1.
  Interventions: Biological: mRNA-1273.351
- mRNA 1273.351 50 ug (Part C) (Experimental): Part C: Participants will receive 1 IM booster dose of 50 ug of mRNA 1273.351 on Day 1.
  Interventions: Biological: mRNA-1273.351
- mRNA-1273/mRNA-1273.351 mixture (Part C) (Experimental): Part C: Participants will receive 1 IM booster dose of 50 ug of mRNA-1273/mRNA-1273.351 mixture on Day 1.
  Interventions: Biological: Biological: mRNA-1273; Biological: mRNA-1273.351

INTERVENTIONS:
Biological: Biological: mRNA-1273 — Sterile liquid for injection
  Arms: Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 18-54 years; Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 55+ years; mRNA-1273/mRNA-1273.351 mixture (Part C); mRNA-1273: Dose 100 ug - Participants Aged 18-54 years; mRNA-1273: Dose 100 ug - Participants Aged 55+ years; mRNA-1273: Dose 50 microgram (ug) - Participants Aged 18-54 years; mRNA-1273: Dose 50 ug - Participants Aged 55+ years
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 18-54 years; Placebo (Part A) and mRNA-1273 100 ug (Part B) - Participants Aged 55+ years
Biological: mRNA-1273.351 — Sterile liquid for injection
  Arms: mRNA 1273.351 20 ug (Part C); mRNA 1273.351 50 ug (Part C); mRNA-1273/mRNA-1273.351 mixture (Part C)

SUMMARY:
This clinical study will assess the safety, reactogenicity, and immunogenicity of 2 dose levels of mRNA-1273 Severe Acute Respiratory Syndrome coronavirus (SARS-COV-2) vaccine in adults 18 years of age or older.

DETAILED DESCRIPTION:
This is a 3-part Phase 2a study, with Part A (Blinded Phase), Part B (Open-label Interventional Phase), and Part C (Rollover Proof of Concept).

Participants in Part A are blinded to their treatment assignment, with participants receiving either 2 active mRNA-1273 vaccine doses or placebo. Part B of the study is designed to offer participants to be unblinded so that participants who received placebo in Part A can request 2 doses of open-label mRNA-1273 vaccine. Additionally, participants who originally received 1 or 2 doses of mRNA-1273 (50 microgram [μg] or 100 μg vaccine) during Part A, will have the opportunity to request to receive a single booster dose of mRNA-1273.

Part C will be a proof-of-concept rollover study to evaluate a vaccine to treat mutations of SARS-CoV2, such as the S-protein of the B.1.351 variant. Part C will include approximately 60 participants, who are currently enrolled in Moderna's Phase 3 mRNA-1273-P301 study (NCT04470427), have already been unblinded, and have previously received 2 doses of mRNA-1273 at least 6 months earlier. At enrollment into Part C of this study, their participation in mRNA-1273-P301 study will be terminated. Part C will evaluate the safety and immunogenicity of 2 dose levels (20 µg and 50 µg) of mRNA-1273.351 and mRNA-1273/mRNA-1273.351 mixture (50 µg total), given as a single booster dose.

ELIGIBILITY:
Key Inclusion Criteria:

Each participant must meet all of the following criteria during the screening period and at Day 1, unless noted otherwise, to be enrolled in this study:

1. Male or female, 18 years of age or older at the time of consent (Screening Visit, Day 0). For Part B, participants must have been previously enrolled in the mRNA-1273 P201 study.
2. Understands and agrees to comply with the study procedures and provides written informed consent.
3. According to the assessment of the investigator, is in good general health and can comply with study procedures.
4. Female participants of nonchildbearing potential may be enrolled in the study. Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening (Day 0) without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the investigator to confirm postmenopausal status.
5. Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

   * Has a negative pregnancy test at Screening (Day 0) and on the day of the first injection (Day 1).
   * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection (Day 1).
   * Has agreed to continue adequate contraception through 3 months following the second injection (Day 29).
   * Is not currently breastfeeding.

   Adequate female contraception is defined as consistent and correct use of a Food and Drug Administration (FDA) approved contraceptive method in accordance with the product label. For example:
   * Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide
   * Intrauterine device
   * Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch), subdermal, or IM route
   * Sterilization of a female participant's monogamous male partner prior to entry into the study Note: periodic abstinence (for example, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
6. Male participants engaging in activity that could result in pregnancy of sexual partners must agree to practice adequate contraception from the time of the first injection and through 3 months after the last injection.

Adequate contraception for male participants is defined as:

* Monogamous relationship with a female partner using an intrauterine device or hormonal contraception (described above)
* Use of barrier methods and spermicide
* History of surgical sterilization
* Male participants with partners who have become pregnant prior to Screening are eligible to participate in the study.

Additional Key Inclusion Criteria for Part C

1. Participants must have been previously enrolled in the mRNA-1273-P301 study and must have received 2 doses of mRNA-1273 in Part A, has been unblinded and aware of their actual treatment in Study mRNA-1273-P301, must have been compliant in Study mRNA-1273-P301 (was not withdrawn or discontinued early), and has been at least 6 months since their second dose in Study mRNA-1273-P301 prior to enrollment in this part.

Key Exclusion Criteria:

Participants meeting any of the following criteria at the Screening Visit (Day 0) or at Day 1, unless noted otherwise, will be excluded from the study:

1. Pregnant or breastfeeding.
2. Is acutely ill or febrile 24 hours prior to or at the Screening Visit (Day 0). Fever is defined as a body temperature ≥38.0°Celsius/100.4°Fahrenheit. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
3. Current treatment with investigational agents for prophylaxis against COVID-19.
4. Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
5. Is a healthcare worker or a member of an emergency response team.
6. Current use of any inhaled substance (for example, tobacco or cannabis smoke, nicotine vapors).
7. History of chronic smoking (≥1 cigarette a day) within 1 year of the Screening Visit (Day 0).
8. History of illegal substance use or alcohol abuse within the past 2 years. This exclusion does not apply to historical cannabis use that was formerly illegal in the participant's state but is legal at the time of Screening.
9. Known history of hypertension, or systolic blood pressure >150 millimeter of mercury (mmHg) in participants in Cohort 1 (≥18 to <55 years old) or systolic blood pressure >160 mmHg in participants in Cohort 2 (≥55 years old) at the Screening Visit (Day 0).
10. Known history of hypotension or systolic blood pressure <85 mmHg at the Screening Visit (Day 0).
11. Diabetes mellitus
12. Diagnosis of chronic pulmonary disease (for example, chronic obstructive pulmonary disease, asthma)
13. Chronic cardiovascular disease
14. Resides in a nursing home
15. Grade 1 or higher toxicity on clinical safety laboratory testing at the Screening Visit (Day 0)
16. Current or previous diagnosis of immunocompromising condition, immune-mediated disease, or other immunosuppressive condition.
17. Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the Screening Visit (Day 0) (for corticosteroids ≥20 milligrams (mg)/day of prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to the Screening Visit (Day 0).
18. Anticipating the need for immunosuppressive treatment at any time during participation in the study.
19. Positive serology for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) type 1 or 2 antibodies identified at the Screening Visit (Day 0).
20. History of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine.
21. Bleeding disorder considered a contraindication to IM injection or phlebotomy.
22. Diagnosis of malignancy within previous 10 years (excluding non-melanoma skin cancer).
23. Has received or plans to receive a licensed vaccine ≤28 days prior to the first injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after any study injection. Licensed influenza vaccines may be received more than 14 days before or after any study injection.
24. Receipt of systemic immunoglobulins or blood products within 3 months prior to the Screening Visit (Day 0) or plans for receipt during the study.
25. Has donated ≥450 mL of blood products within 28 days prior to the Screening Visit (Day 0) or plans to donate blood products during the study.
26. Participated in an interventional clinical study (other than mRNA-1273 P301) within 28 days prior to the Screening Visit (Day 0) or plans to do so while participating in this study.
27. Is an immediate family member or household member of study personnel

Additional Key Exclusion Criteria for Part C

1. Is SARS-CoV-2 positive by Reverse transcription polymerase chain reaction (RT-PCR) (central or local testing) at baseline or at any time during the mRNA-1273-P301 study regardless of the presence or absence of symptoms consistent with COVID-19.
2. Had any SAE in the mRNA-1273-P301 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Meridian Clinical Research, Savannah, Georgia
  - Alliance for Multispecialty Research, Newton, Kansas
  - Alliance for Multispecialty Research, Kansas City, Missouri
  - Meridian Clinical Research, Norfolk, Nebraska
  - Trial Management Associates, Wilmington, North Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Benchmark Research, Austin, Texas
  - Benchmark Research, San Angelo, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirste I, Hortsch S, Grunert VP, Legault H, Maglinao M, Eichenlaub U, Kashlan B, Pajon R, Jochum S. Quantifying the Vaccine-Induced Humoral Immune Response to Spike-Receptor Binding Domain as a Surrogate for Neutralization Testing Following mRNA-1273 (Spikevax) Vaccination Against COVID-19. Infect Dis Ther. 2023 Jan;12(1):177-191. doi: 10.1007/s40121-022-00711-y. Epub 2022 Nov 15. PMID 36376733
- [Derived] Chalkias S, Eder F, Essink B, Khetan S, Nestorova B, Feng J, Chen X, Chang Y, Zhou H, Montefiori D, Edwards DK, Girard B, Pajon R, Dutko FJ, Leav B, Walsh SR, Baden LR, Miller JM, Das R. Safety, immunogenicity and antibody persistence of a bivalent Beta-containing booster vaccine against COVID-19: a phase 2/3 trial. Nat Med. 2022 Nov;28(11):2388-2397. doi: 10.1038/s41591-022-02031-7. Epub 2022 Oct 6. PMID 36202997
- [Derived] Chu L, Vrbicky K, Montefiori D, Huang W, Nestorova B, Chang Y, Carfi A, Edwards DK, Oestreicher J, Legault H, Dutko FJ, Girard B, Pajon R, Miller JM, Das R, Leav B, McPhee R. Immune response to SARS-CoV-2 after a booster of mRNA-1273: an open-label phase 2 trial. Nat Med. 2022 May;28(5):1042-1049. doi: 10.1038/s41591-022-01739-w. Epub 2022 Mar 3. PMID 35241844
- [Derived] Choi A, Koch M, Wu K, Chu L, Ma L, Hill A, Nunna N, Huang W, Oestreicher J, Colpitts T, Bennett H, Legault H, Paila Y, Nestorova B, Ding B, Montefiori D, Pajon R, Miller JM, Leav B, Carfi A, McPhee R, Edwards DK. Safety and immunogenicity of SARS-CoV-2 variant mRNA vaccine boosters in healthy adults: an interim analysis. Nat Med. 2021 Nov;27(11):2025-2031. doi: 10.1038/s41591-021-01527-y. Epub 2021 Sep 15. PMID 34526698
- [Derived] Chu L, McPhee R, Huang W, Bennett H, Pajon R, Nestorova B, Leav B; mRNA-1273 Study Group. A preliminary report of a randomized controlled phase 2 trial of the safety and immunogenicity of mRNA-1273 SARS-CoV-2 vaccine. Vaccine. 2021 May 12;39(20):2791-2799. doi: 10.1016/j.vaccine.2021.02.007. Epub 2021 Feb 9. PMID 33707061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in Part A were blinded to study treatment. After completion of Part A, participants could have chosen to be unblinded and to participate in Part B (open-label). Participants in Part C (proof-of-concept rollover) were unblinded and had received 2 doses of mRNA-1273 in Study mRNA-1273-P301 (Study P301; NCT04470427).
Pre-assignment Details: Part A participants received 50 microgram (µg) mRNA-1273, 100 µg mRNA-1273, or placebo (N=600). Participants who received placebo in Part A, received 100 ug mRNA-1273 in Part B (N=158). Participants who received 50 or 100 ug mRNA-1273 in Part A, received 50 ug mRNA-1273 in Part B (N=344). Participants in Part C (N=60) received a booster dose of 20 or 50 µg of mRNA-1273.351 or 50 µg mRNA-1273/mRNA-1273.351 mixture. Total number of enrolled participants for the study=660.
Groups:
- Part A: 50 ug mRNA-1273: Participants received 1 intramuscular (IM) injection of 50 ug mRNA-1273 on Day 1 and on Day 29.
- Part A: 100 ug mRNA-1273: Participants received 1 IM injection of 100 ug mRNA-1273 on Day 1 and on Day 29.
- Part A: Placebo: Participants received 1 IM injection of mRNA-1273-matching placebo on Day 1 and on Day 29.
- Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273: Participants who chose to be unblinded and received 50 ug mRNA-1273 during Part A, received 1 IM injection of 50 ug mRNA-1273 during Part B.
- Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273: Participants who chose to be unblinded and received 100 ug mRNA-1273 during Part A, received 1 IM injection of 50 ug mRNA-1273 during Part B.
- Part B: Placebo Then 100 ug mRNA-1273: Participants who chose to be unblinded and received mRNA-1273-matching placebo during Part A, received 2 IM injections of 100 ug mRNA-1273 28 days apart during Part B.
- Part C: 20 ug mRNA-1273.351: Participants received 1 IM injection of 20 ug mRNA-1273.351 (booster dose) on Day 1.
- Part C: 50 ug mRNA-1273.351: Participants received 1 IM injection of 50 ug mRNA-1273.351 (booster dose) on Day 1.
- Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture: Participants received 1 IM injection of 50 ug mRNA-1273/mRNA-1273.351 mixture (booster dose) on Day 1.
Period: Part A (Blinded Phase)
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Started | 200 | 200 | 200 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug During Part A | 200 | 200 | 200 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 188 | 185 | 182 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 15 | 18 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent (COVID-19 non-infection related) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent (other) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other than Specified | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Open-Label Interventional Phase)
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Started | 0 | 0 | 0 | 173 | 171 | 158 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug During Part B | 0 | 0 | 0 | 173 | 171 | 158 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 161 | 166 | 152 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 12 | 5 | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 1 | 4 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 6 | 3 | 2 | 0 | 0 | 0
Period: Part C (Rollover Proof of Concept)
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Started | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Not completed — Withdrawal of consent (other) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: All participants who received any study injection in their respective part of the study. Note, participants who received placebo in Part A, received 100 ug mRNA-1273 in Part B (N=158). Participants who received 50 or 100 ug mRNA-1273 in Part A, received 50 ug mRNA-1273 in Part B (N=344). Since Baseline Characteristics data for participants in Part B are included in Part A, separate columns are not reported here for Part B.
Groups:
- Part A: 50 ug mRNA-1273: Participants received 1 IM injection of 50 ug mRNA-1273 on Day 1 and on Day 29.
- Total: Total of all reporting groups
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture | Total
Number analyzed (Participants) | 200 | 200 | 200 | 20 | 20 | 20 | 660
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 55 years | 100 | 100 | 100 | 13 | 9 | 9 | 331
  >=55 years | 100 | 100 | 100 | 7 | 11 | 11 | 329
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 124 | 129 | 15 | 9 | 8 | 422
  Male | 63 | 76 | 71 | 5 | 11 | 12 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 16 | 1 | 0 | 1 | 49
  Not Hispanic or Latino | 184 | 184 | 184 | 19 | 20 | 19 | 610
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 188 | 188 | 193 | 20 | 19 | 19 | 627
  Black or African American | 5 | 8 | 3 | 0 | 0 | 0 | 16
  Asian | 2 | 2 | 3 | 0 | 1 | 0 | 8
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Multiracial | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Other | 1 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs, including local and systemic ARs were collected in the eDiary. Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. All solicited ARs (local and systemic) considered causally related to injection. ARs were graded 0-4 as reviewed and confirmed by Investigator; lower score indicates lower severity and a higher score indicates greater severity. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set for Parts A, B, and C included all participants who received any study injection in the applicable part of the study and contributed any solicited AR data (that is, had at least 1 post-baseline solicited safety assessment in the applicable part of the study). Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 200 | 200 | 200 | 164 | 167 | 157 | 19 | 19 | 20
Participants
  Grade 1 | 95 | 69 | 72 | 65 | 73 | 50 | 13 | 10 | 12
  Grade 2 | 61 | 90 | 21 | 59 | 59 | 71 | 6 | 2 | 3
  Grade 3 | 25 | 32 | 6 | 29 | 18 | 28 | 0 | 2 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent AE (TEAE) was defined as any event not present before exposure to vaccine or any event already present that worsens in intensity or frequency after exposure. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsens from baseline and is considered clinically significant in the medical and scientific judgment of the Investigator. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Month 15), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set: All participants who received any study injection in their respective part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 200 | 200 | 200 | 173 | 171 | 158 | 20 | 20 | 20
Participants | 57 | 56 | 51 | 17 | 25 | 42 | 3 | 3 | 4

3. Primary Outcome: Number of Participants With Medically-Attended Adverse Events (MAAEs)
Description: An MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner (HCP). A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Month 15
Population: Safety Set: All participants who received any study injection in their respective part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 200 | 200 | 200 | 173 | 171 | 158 | 20 | 20 | 20
Participants | 74 | 38 | 64 | 42 | 47 | 59 | 7 | 3 | 7

4. Primary Outcome: Number of Participants With SAEs
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Month 15
Population: Safety Set: All participants who received any study injection in their respective part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 200 | 200 | 200 | 173 | 171 | 158 | 20 | 20 | 20
Participants | 5 | 2 | 0 | 2 | 2 | 2 | 0 | 1 | 0

5. Primary Outcome: Part A: Level of Severe Acute Respiratory Syndrome Coronavirus (SARS-COV-2)-Specific Binding Antibody (bAb) as Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: The geometric mean (GM) level of VAC58 spike immunoglobulin G (IgG) antibodies, as measured by ELISA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values that were greater than the upper limit of quantification (ULOQ) were converted to the ULOQ if actual values were not available. LLOQ was 1 and ULOQ was 2052. The 95% confidence intervals (CIs) were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM value, respectively, then back transformed to the original scale for presentation.
Time Frame: Days 1 (Baseline), 29, 43, 57, and 209
Population: Per-Protocol (PP) Set included randomized participants who received any study injection, had required baseline (Day 1) data, had ≥1 post-injection assessment for the analysis endpoint, complied with injection schedule, had post-injection results available for ≥1 assay component corresponding to immunogenicity analysis, did not have SARS-CoV-2 infection, and had no major protocol deviations impacting applicable immune response. Number Analyzed = participants evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units per mL (AU/mL)
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo
Number analyzed (Participants) | 185 | 189 | 186
arbitrary units per mL (AU/mL)
  Day 1 (Baseline) | 0.70 [0.63 to 0.78] | 0.67 [0.60 to 0.73] | 0.67 [0.61 to 0.73]
  Day 29: number analyzed (Participants) | 183 | 189 | 182
  Day 29 | 59.42 [52.05 to 67.82] | 81.51 [70.19 to 94.67] | 0.68 [0.61 to 0.76]
  Day 43: number analyzed (Participants) | 176 | 180 | 180
  Day 43 | 720.85 [660.30 to 786.96] | 834.66 [765.28 to 910.33] | 0.65 [0.59 to 0.71]
  Day 57: number analyzed (Participants) | 176 | 174 | 174
  Day 57 | 519.48 [474.00 to 569.33] | 647.22 [588.98 to 711.21] | 0.67 [0.60 to 0.75]
  Day 209: number analyzed (Participants) | 170 | 174 | 154
  Day 209 | 97.02 [87.58 to 107.47] | 128.00 [114.44 to 143.18] | 0.91 [0.73 to 1.14]

6. Primary Outcome: Part B: Level of SARS-CoV-2-Specific bAb as Measured by ELISA
Description: The GM level of VAC65 spike IgG antibodies, as measured by ELISA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ are converted to the ULOQ. LLOQ was 1 and ULOQ was 2052. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM value, respectively, then back transformed to the original scale for presentation. The PP Set included participants with a study injection, required baseline data, had postinjection results at timepoint of primary interest for immunogenicity analysis, no major protocol deviations impacting immune response, and didn't have SARS-CoV-2.
Time Frame: Days 1 (Baseline) and 29
Population: PP Set. Number Analyzed=participants evaluable at specified timepoint. Immunogenicity samples from the "Part B: Placebo then 100 ug mRNA" arm were not tested and no data were generated as results were not thought to provide additional information. After Part B samples were obtained, it was determined that the extensive results for immunogenicity profiles of 2 doses of 100 ug mRNA-1273 that were obtained during Part A of this study and in Study P301 demonstrated enough immune response data.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273
Number analyzed (Participants) | 146 | 149
AU/mL
  Day 1 (Baseline): number analyzed (Participants) | 145 | 147
  Day 1 (Baseline) | 86.29 [76.89 to 96.83] | 109.56 [96.79 to 124.02]
  Day 29: number analyzed (Participants) | 143 | 149
  Day 29 | 1069.73 [992.92 to 1152.49] | 1083.21 [1018.75 to 1151.75]

7. Secondary Outcome: Part A: Titer of SARS-CoV-2-Specific Neutralizing Antibody (nAb)
Description: The GM titer (microneutralization [MN] and MN50) of serum nAb against SARS-CoV-2 as measured by live virus MN assays is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. For MN, LLOQ was 40 and ULOQ was 1280 at Days 1 (Baseline), 29, 43, and 57. For MN50, LLOQ was 91.10 and ULOQ was 2031.87 at Days 1 (Baseline), 29, 43, and 57. For MN, LLOQ was 160 and ULOQ was 1280 at Day 209. For MN50, LLOQ was 318.46 and ULOQ was 1917.83 at Day 209. The 95% CI was calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM titer, then back transformed to the original scale for presentation.
Time Frame: Days 1 (Baseline), 29, 43, 57, and 209
Population: PP Set included randomized participants who received any study injection, had required baseline (Day 1) data, had ≥1 post-injection assessment for the analysis endpoint, complied with injection schedule, had post-injection results available for ≥1 assay component corresponding to immunogenicity analysis, did not have SARS-CoV-2 infection, and had no major protocol deviations impacting applicable immune response. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo
Number analyzed (Participants) | 185 | 189 | 186
titers
  MN, Day 1 (Baseline) | 20.6 [20.0 to 21.2] | 20.6 [19.7 to 21.5] | 20.8 [20.1 to 21.4]
  MN, Day 29: number analyzed (Participants) | 184 | 187 | 184
  MN, Day 29 | 112.2 [94.9 to 132.7] | 149.6 [127.3 to 175.9] | 21.9 [20.5 to 23.5]
  MN, Day 43: number analyzed (Participants) | 174 | 181 | 180
  MN, Day 43 | 1145.4 [1101.3 to 1191.1] | 1185.8 [1142.9 to 1230.3] | 21.2 [20.1 to 22.4]
  MN, Day 57: number analyzed (Participants) | 176 | 177 | 175
  MN, Day 57 | 1090.6 [1038.9 to 1144.9] | 1095.5 [1041.5 to 1152.2] | 21.8 [20.4 to 23.4]
  MN, Day 209: number analyzed (Participants) | 171 | 174 | 153
  MN, Day 209 | 254.4 [219.4 to 294.9] | 354.8 [309.2 to 407.2] | 85.3 [80.6 to 90.2]
  MN50, Day 1 (Baseline) | 46.500 [45.425 to 47.600] | 46.684 [44.957 to 48.477] | 47.109 [45.745 to 48.512]
  MN50, Day 29: number analyzed (Participants) | 184 | 187 | 184
  MN50, Day 29 | 173.750 [148.550 to 203.225] | 227.433 [194.207 to 266.343] | 49.231 [46.355 to 52.285]
  MN50, Day 43: number analyzed (Participants) | 174 | 181 | 180
  MN50, Day 43 | 1761.660 [1690.216 to 1836.124] | 1813.480 [1741.280 to 1888.673] | 48.059 [45.820 to 50.408]
  MN50, Day 57: number analyzed (Participants) | 176 | 177 | 175
  MN50, Day 57 | 1632.442 [1550.245 to 1718.998] | 1656.064 [1570.464 to 1746.330] | 49.141 [46.267 to 52.194]
  MN50, Day 209: number analyzed (Participants) | 171 | 174 | 153
  MN50, Day 209 | 401.508 [350.667 to 459.720] | 538.798 [472.772 to 614.045] | 167.002 [159.249 to 175.133]

8. Secondary Outcome: Part B: Titer of SARS-CoV-2-Specific nAb
Description: The GM titer (50% inhibitory dose [ID50], 80% inhibitory dose [ID80]) of nAb against SARS-CoV-2 pseudotyped viruses as measured by pseudovirus nAb assay is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were converted to the ULOQ if actual values were not available. LLOQ was 18.5 and ULOQ was 45118 for IC50. LLOQ was 14.3 and ULOQ was 10232 for ID80. The 95% CI was calculated based on the t-distribution of the log-transformed values for GM titer, then back transformed to the original scale for presentation. The PP Set included participants with a study injection, required baseline data, had postinjection results at timepoint of primary interest for immunogenicity analysis, no major protocol deviations impacting immune response, and didn't have SARS-CoV-2.
Time Frame: Days 1 (Baseline), 29, and 181
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273
Number analyzed (Participants) | 146 | 149
titers
  ID50, Day 1 (Baseline): number analyzed (Participants) | 145 | 149
  ID50, Day 1 (Baseline) | 104.658 [88.282 to 124.070] | 150.224 [125.726 to 179.495]
  ID50, Day 29 | 1834.309 [1600.233 to 2102.623] | 1951.735 [1729.606 to 2202.392]
  ID50, Day 181: number analyzed (Participants) | 38 | 147
  ID50, Day 181 | 915.331 [622.504 to 1345.904] | 673.273 [578.167 to 784.025]
  ID80, Day 1 (Baseline): number analyzed (Participants) | 145 | 149
  ID80, Day 1 (Baseline) | 39.646 [33.789 to 46.518] | 55.686 [47.459 to 65.341]
  ID80, Day 29 | 696.085 [609.203 to 795.358] | 736.617 [661.040 to 820.835]
  ID80, Day 181: number analyzed (Participants) | 38 | 147
  ID80, Day 181 | 291.791 [203.597 to 418.189] | 228.635 [197.044 to 265.291]

9. Secondary Outcome: Part C: Titer of SARS-CoV-2-Specific nAb
Description: The GM titer (ID50, ID80) of nAb against SARS-CoV-2 pseudotyped viruses (original strain and beta variant [B.1.351]) as measured by pseudovirus nAb assay is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were converted to the ULOQ if actual values were not available. For NAb ID50 Titers, LLOQ was 18.5 and ULOQ was 45118. For NAb ID80 Titers, LLOQ was 14.3 and ULOQ was 10232. For NAb ID50 Titers against B.1.351, LLOQ was 19.5 and ULOQ was 385.7. For NAb ID80 Titers against B.1.351, LLOQ was 12.5 and ULOQ was 102.2. The 95% CI was calculated based on the t-distribution of the log-transformed values for GM titer, then back transformed to the original scale for presentation.
Time Frame: Days 1 (Baseline), 8, 15, 29, and 181
Population: PP Set included participants who received any study injection, had required baseline (Day 1) data, had ≥1 post-injection assessment for the analysis endpoint, complied with injection schedule, had post-injection results available for ≥1 assay component corresponding to immunogenicity analysis, did not have SARS-CoV-2 infection, and had no major protocol deviations impacting applicable immune response. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 19 | 20 | 20
titers
  ID50 Against Original Strain, Day 1 (Baseline) | 196.107 [133.338 to 288.424] | 156.011 [80.546 to 302.180] | 79.572 [53.625 to 118.074]
  ID50 Against Original Strain, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID50 Against Original Strain, Day 8 | 1089.901 [748.146 to 1587.770] | 1568.894 [1030.722 to 2388.062] | 1183.096 [900.313 to 1554.700]
  ID50 Against Original Strain, Day 15 | 2221.382 [1434.353 to 3440.255] | 1725.415 [1212.131 to 2456.053] | 3082.946 [1891.502 to 5024.874]
  ID50 Against Original Strain, Day 29 | 1808.133 [1323.211 to 2470.767] | 1757.179 [1117.782 to 2762.324] | 3691.896 [2330.908 to 5847.548]
  ID50 Against Original Strain, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID50 Against Original Strain, Day 181 |  | 512.129 [303.261 to 864.853] |
  ID80 Against Original Strain, Day 1 (Baseline) | 76.279 [53.035 to 109.712] | 56.344 [33.804 to 93.911] | 30.774 [21.565 to 43.915]
  ID80 Against Original Strain, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID80 Against Original Strain, Day 8 | 448.109 [300.430 to 668.381] | 500.158 [341.180 to 733.214] | 458.435 [351.348 to 598.161]
  ID80 Against Original Strain, Day 15 | 730.018 [509.454 to 1046.073] | 678.926 [462.561 to 996.498] | 947.774 [647.781 to 1386.696]
  ID80 Against Original Strain, Day 29 | 632.263 [460.549 to 868.001] | 615.967 [397.103 to 955.460] | 1156.267 [743.617 to 1797.907]
  ID80 Against Original Strain, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID80 Against Original Strain, Day 181 |  | 182.837 [108.300 to 308.673] |
  ID50 Against B.1.351, Day 1 (Baseline) | 45.574 [28.832 to 72.036] | 32.026 [19.758 to 51.911] | 18.338 [13.572 to 24.776]
  ID50 Against B.1.351, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID50 Against B.1.351, Day 8 | 919.281 [592.738 to 1425.720] | 1088.511 [670.315 to 1767.610] | 706.141 [456.010 to 1093.475]
  ID50 Against B.1.351, Day 15 | 1088.432 [736.353 to 1608.854] | 1113.392 [652.885 to 1898.716] | 1166.830 [760.230 to 1790.895]
  ID50 Against B.1.351, Day 29 | 1537.029 [1066.352 to 2215.458] | 1116.885 [714.119 to 1746.813] | 1129.955 [742.454 to 1719.699]
  ID50 Against B.1.351, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID50 Against B.1.351, Day 181 |  | 141.773 [76.471 to 262.839] |
  ID80 Against B.1.351, Day 1 (Baseline) | 17.403 [10.870 to 27.863] | 15.046 [10.088 to 22.442] | 8.326 [6.727 to 10.306]
  ID80 Against B.1.351, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID80 Against B.1.351, Day 8 | 289.360 [196.260 to 426.626] | 313.644 [203.582 to 483.210] | 225.475 [160.419 to 316.915]
  ID80 Against B.1.351, Day 15 | 435.078 [300.742 to 629.418] | 371.579 [228.889 to 603.223] | 413.424 [284.856 to 600.020]
  ID80 Against B.1.351, Day 29 | 486.398 [341.630 to 692.511] | 345.827 [214.472 to 557.633] | 362.540 [249.138 to 527.560]
  ID80 Against B.1.351, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID80 Against B.1.351, Day 181 |  | 55.887 [29.969 to 104.220] |

10. Secondary Outcome: Part A: Percentage of Participants With Seroconversion From Baseline
Description: Based on MN titers and MN50 titers of serum nAb against SARS-CoV-2 as measured by live virus MN assays, percentage of participants with seroconversion from baseline are reported with 2-sided 95% CI using the Clopper-Pearson method at each post-baseline timepoint. Seroconversion at a participant level was defined as a change of nAb titer from below the limit of detection (LOD) or LLOQ to equal to or above LOD or LLOQ (respectively), or a 4-times or higher titer ratio in participants with pre-existing nAb titers. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. For MN, LLOQ was 40 and ULOQ was 1280. For MN50, LLOQ was 91.10 and ULOQ was 2031.87.
Time Frame: Days 29, 43, and 57
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo
Number analyzed (Participants) | 168 | 180 | 178
percentage of participants
  MN Titer, Day 29 | 78.0 [70.9 to 84.0] | 88.9 [83.4 to 93.1] | 1.7 [0.3 to 4.8]
  MN Titer, Day 43: number analyzed (Participants) | 141 | 150 | 175
  MN Titer, Day 43 | 100 [97.4 to 100.0] | 100 [97.6 to 100.0] | 0.6 [0.0 to 3.1]
  MN Titer, Day 57: number analyzed (Participants) | 150 | 152 | 171
  MN Titer, Day 57 | 100 [97.6 to 100.0] | 100 [97.6 to 100.0] | 1.8 [0.4 to 5.0]
  MN50 Titer, Day 29 | 65.5 [57.8 to 72.6] | 76.7 [69.8 to 82.6] | 1.1 [0.1 to 4.0]
  MN50 Titer, Day 43: number analyzed (Participants) | 141 | 150 | 175
  MN50 Titer, Day 43 | 100 [97.4 to 100.0] | 100 [97.6 to 100.0] | 0.6 [0.0 to 3.1]
  MN50 Titer, Day 57: number analyzed (Participants) | 150 | 152 | 171
  MN50 Titer, Day 57 | 100 [97.6 to 100.0] | 100 [97.6 to 100.0] | 1.8 [0.4 to 5.0]

11. Secondary Outcome: Part B: Percentage of Participants With Seroconversion From Baseline
Description: Based on ID50 and ID80 titers of nAb against SARS-CoV-2 pseudotyped viruses as measured by pseudovirus nAb assay, % of participants with seroconversion from baseline reported with 2-sided 95% CI using Clopper-Pearson method at each postbaseline timepoint. Seroconversion at participant level defined as change of nAb titer from below LOD or LLOQ to equal to or above LOD or LLOQ (respectively) or 4-times or higher titer ratio in participants with preexisting nAb titers. Antibody values <LLOQ replaced by 0.5*LLOQ. Values >ULOQ converted to ULOQ. LLOQ: 18.5 and ULOQ: 45118 for IC50. LLOQ: 14.3 and ULOQ: 10232 for ID80. 95% CI calculated based on t-distribution of log-transformed values for GMT, then back transformed to original scale for presentation. PP Set: participants with a study injection, required baseline data, had postinjection results at timepoint of primary interest for immunogenicity analysis, no major protocol deviations impacting immune response, and didn't have SARS-CoV-2.
Time Frame: Days 29 and 181
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273
Number analyzed (Participants) | 146 | 149
percentage of participants
  ID50, Day 29 | 92.4 [86.8 to 96.2] | 87.9 [81.6 to 92.7]
  ID50, Day 181: number analyzed (Participants) | 38 | 147
  ID50, Day 181 | 81.6 [65.7 to 92.3] | 54.4 [46.0 to 62.6]
  ID80, Day 29 | 95.2 [90.3 to 98.0] | 93.3 [88.0 to 96.7]
  ID80, Day 181: number analyzed (Participants) | 38 | 147
  ID80, Day 181 | 78.9 [62.7 to 90.4] | 53.7 [45.3 to 62.0]

12. Secondary Outcome: Part C: Percentage of Participants With Seroconversion From Baseline
Description: Based on ID50 titers and ID80 titers of nAb against SARS-CoV-2 pseudotyped viruses (original strain and beta variant [B.1.351]) as measured by pseudovirus nAb assay, percentage of participants with seroconversion from baseline are reported with 2-sided 95% CI using Clopper-Pearson method at each post-baseline timepoint. Seroconversion at participant level defined as a change of nAb titer from below LOD or LLOQ ≥LOD or LLOQ (respectively), or a 4-times or higher titer ratio in participants with pre-existing nAb titers. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values >ULOQ were converted to ULOQ. NAb ID50 Titers: LLOQ was 18.5 and ULOQ was 45118. NAb ID80 Titers: LLOQ was 14.3 and ULOQ was 10232. NAb ID50 Titers against B.1.351: LLOQ was 19.5 and ULOQ was 385.7. NAb ID80 Titers against B.1.351: LLOQ was 12.5 and ULOQ was 102.2. 95% CI calculated based on t-distribution of log-transformed values for GMT, then back transformed to original scale for presentation.
Time Frame: Days 8, 15, 29, and 181
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 19 | 20 | 20
percentage of participants
  ID50 Against Original Strain, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID50 Against Original Strain, Day 8 | 47.4 [24.4 to 71.1] | 78.9 [54.4 to 93.9] | 100 [83.2 to 100.0]
  ID50 Against Original Strain, Day 15 | 78.9 [54.4 to 93.9] | 90.0 [68.3 to 98.8] | 95.0 [75.1 to 99.9]
  ID50 Against Original Strain, Day 29 | 84.2 [60.4 to 96.6] | 95.0 [75.1 to 99.9] | 100 [83.2 to 100.0]
  ID50 Against Original Strain, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID50 Against Original Strain, Day 181 |  | 38.9 [17.3 to 64.3] |
  ID80 Against Original Strain, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID80 Against Original Strain, Day 8 | 68.4 [43.4 to 87.4] | 84.2 [60.4 to 96.6] | 95.0 [75.1 to 99.9]
  ID80 Against Original Strain, Day 15 | 84.2 [60.4 to 96.6] | 95.0 [75.1 to 99.9] | 100 [83.2 to 100.0]
  ID80 Against Original Strain, Day 29 | 84.2 [60.4 to 96.6] | 95.0 [75.1 to 99.9] | 95.0 [75.1 to 99.9]
  ID80 Against Original Strain, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID80 Against Original Strain, Day 181 |  | 38.9 [17.3 to 64.3] |
  ID50 Against B.1.351, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID50 Against B.1.351, Day 8 | 100 [82.4 to 100.0] | 100 [82.4 to 100.0] | 100 [83.2 to 100.0]
  ID50 Against B.1.351, Day 15 | 94.7 [74.0 to 99.9] | 100 [83.2 to 100.0] | 100 [83.2 to 100.0]
  ID50 Against B.1.351, Day 29 | 100 [82.4 to 100.0] | 100 [83.2 to 100.0] | 100 [83.2 to 100.0]
  ID50 Against B.1.351, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID50 Against B.1.351, Day 181 |  | 61.1 [35.7 to 82.7] |
  ID80 Against B.1.351, Day 8: number analyzed (Participants) | 19 | 19 | 20
  ID80 Against B.1.351, Day 8 | 94.7 [74.0 to 99.9] | 94.7 [74.0 to 99.9] | 100 [83.2 to 100.0]
  ID80 Against B.1.351, Day 15 | 94.7 [74.0 to 99.9] | 100 [83.2 to 100.0] | 100 [83.2 to 100.0]
  ID80 Against B.1.351, Day 29 | 100 [82.4 to 100.0] | 100 [83.2 to 100.0] | 100 [83.2 to 100.0]
  ID80 Against B.1.351, Day 181: number analyzed (Participants) | 0 | 18 | 0
  ID80 Against B.1.351, Day 181 |  | 55.6 [30.8 to 78.5] |

13. Primary Outcome: Part C: Level of SARS-CoV-2-Specific bAb as Measured by MSD
Description: The GM level of SARS-CoV-2 protein antibody against B.1.351, as measured by MSD MULTIPLEX is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ are converted to the ULOQ. LLOQ was 18 and ULOQ was 4200000. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM value, respectively, then back transformed to the original scale for presentation.
Time Frame: Days 1 (Baseline), 8, 15, and 29
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- 50 ug mRNA-1273.351: Participants received 1 IM injection of 50 ug mRNA-1273.351 (booster dose) on Day 1.
Arm/Group | Part C: 20 ug mRNA-1273.351 | 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
Number analyzed (Participants) | 19 | 20 | 20
AU/mL
  Day 1 (Baseline) | 59742.3 [43057.8 to 82891.8] | 44921.5 [28539.6 to 70706.5] | 33409.8 [25264.8 to 44180.6]
  Day 8: number analyzed (Participants) | 19 | 19 | 20
  Day 8 | 240180.0 [166361.1 to 346754.3] | 267002.2 [199939.9 to 356558.2] | 228572.0 [178986.7 to 291894.2]
  Day 15 | 297880.2 [224089.6 to 395969.4] | 418215.3 [311988.7 to 560610.2] | 384521.1 [282461.4 to 523457.3]
  Day 29 | 297962.7 [227337.5 to 390528.5] | 345765.9 [251640.5 to 475098.5] | 367714.1 [268913.2 to 502815.1]

ADVERSE EVENTS:
Time Frame: Up to Month 15
Description: Safety Set: All participants who received any study injection in their respective part of the study. Note, not all solicited ARs were considered AEs. The Investigator reviewed whether the solicited AR was also to be recorded as an AE.
Arm/Group | Part A: 50 ug mRNA-1273 | Part A: 100 ug mRNA-1273 | Part A: Placebo | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 | Part B: Placebo Then 100 ug mRNA-1273 | Part C: 20 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273.351 | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200 | 0/200 | 0/173 | 0/171 | 0/158 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 5/200 | 2/200 | 0/200 | 2/173 | 2/171 | 2/158 | 0/20 | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 105/200 | 76/200 | 94/200 | 51/173 | 62/171 | 70/158 | 8/20 | 4/20 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 50 ug mRNA-1273 (N=200) | Part A: 100 ug mRNA-1273 (N=200) | Part A: Placebo (N=200) | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 (N=173) | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 (N=171) | Part B: Placebo Then 100 ug mRNA-1273 (N=158) | Part C: 20 ug mRNA-1273.351 (N=20) | Part C: 50 ug mRNA-1273.351 (N=20) | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture (N=20)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system cyst (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Struck by lightning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma stage IV (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 50 ug mRNA-1273 (N=200) | Part A: 100 ug mRNA-1273 (N=200) | Part A: Placebo (N=200) | Part B: 50 ug mRNA-1273 Then 50 ug mRNA-1273 (N=173) | Part B: 100 ug mRNA-1273 Then 50 ug mRNA-1273 (N=171) | Part B: Placebo Then 100 ug mRNA-1273 (N=158) | Part C: 20 ug mRNA-1273.351 (N=20) | Part C: 50 ug mRNA-1273.351 (N=20) | Part C: 50 ug mRNA-1273/mRNA-1273.351 Mixture (N=20)
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 4 | 2 | 2 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 2 | 26 | 9 | 8 | 16 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 3 | 0 | 2 | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 3 | 4 | 4 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 2 | 0 | 2 | 2 | 2 | 3 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperoestrogenism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 2 | 3 | 2 | 2 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 16 | 9 | 8 | 3 | 8 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2
Diastolic hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4 | 2 | 3 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 2 | 4 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 3 | 3 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 1 | 2 | 2 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 0 | 4 | 2 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 2 | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 16 | 5 | 7 | 1 | 7 | 5 | 0 | 1 | 1
Injection site pain (General disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Axillary pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hormone level abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Computerised tomogram coronary artery abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulpless tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fascial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT04405076/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04405076/SAP_001.pdf
  • Informed Consent Form (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT04405076/ICF_002.pdf